CLINICAL TRIAL: NCT06436690
Title: Optimizing Antibiotics Prescription: A Stepped-Wedge Randomized Trial
Brief Title: Optimizing Antibiotics Prescription
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Responsible Party: Principal Investigator, Yubraj Acharya, Ph.D., Associate Professor, Penn State University
Allocation: Not Applicable | Model: Crossover | Masking: Double | Purpose: Health Services Research
Other Study IDs: STUDY00025143
Record Dates: First submitted 2024-05-24; First posted 2024-05-31 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Antimicrobial Resistance

STUDY DESIGN:
Intervention Model Description: This is a stepped-wedge randomized controlled trial
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): During this phase, physicians do not receive any intervention.
- Diagnosis Mandate (Experimental): In this phase, physicians receive a refresher training on AMR and a letter requiring the physicians to specify the diagnosis in their prescription note.
  Interventions: Behavioral: Diagnosis Mandate
- Feedback (Experimental): In this phase, physicians receive a customized feedback letter on their prescription behavior, including antibiotics prescription rate.
  Interventions: Behavioral: Individualized Feedback

INTERVENTIONS:
Behavioral: Diagnosis Mandate — The intervention consists of: a) a Refresher Training on AMR, and (b) a Diagnosis Mandate.
  Arms: Diagnosis Mandate
Behavioral: Individualized Feedback — Physicians receive a customized feedback on their prescription behavior, including antibiotics prescription rate.
  Arms: Feedback

SUMMARY:
Interventions that are low-cost, do not add substantially to the physician workload, are consistent with good physician practices and WHO guidelines, and serve as a reminder on the risks of overprescribing antibiotics are critically needed. The overall goal of the proposed project is to test the effect of two behavioral interventions targeted to junior physicians-specifically, requiring them to specify the diagnosis in the prescription note and providing feedback-on their antibiotics prescription rate; examine the intervention's effects across gender and caste; and draw lessons for scaling up the intervention.

DETAILED DESCRIPTION:
Antimicrobial resistance (AMR) is one of the top ten threats to global health. Limited existing evidence from Nepal, the site for the proposed study, suggests that physicians "err on the side of caution" by prescribing antibiotics even for viral conditions, which contributes to AMR. Interventions that are low-cost, do not add substantially to the physician workload, are consistent with good physician practices and WHO guidelines, and serve as a reminder on the risks of overprescribing antibiotics are critically needed. The overall goal of the proposed project is to test the effect of a behavioral intervention targeted to junior physicians-specifically, requiring them to specify the diagnosis in the prescription note and providing feedback-on their antibiotics prescription rate; examine the intervention's effects across gender and caste; and draw lessons for scaling up the intervention.

The specific objectives are the following:

Objective 1. Assess the effect of a behavioral intervention targeted to junior physicians on antibiotics prescription rate, including by caste and gender of the patient. A stepped-wedge randomized control trial (RCT) will be conducted among 60 junior physicians in five hospitals (1 government, 2 private teaching, and 2 community) in Nepal. The intervention will be rolled out sequentially across the hospitals and data will be collected from patients (n=3,600) both before and after the intervention. The intervention will consist of three components: (a) a Refresher Training on AMR, (b) a Diagnosis Mandate, and (c) an Individualized Feedback.

Objective 2. Identify barriers to scaling up the intervention beyond the study's site and strategies for their mitigation. After preliminary analysis of the quantitative data, key informant interviews with national- and provincial- level health policy makers (n=5), and in-depth interviews with physicians (n=5) and hospital managers (n=5) will be conducted.

Objective 3. Assess the extent to which physicians prescribe antibiotics correctly. From a subset of patients (n=120, i.e., 2 per physician), more detailed medical information will be collected and analyzed from their outpatient booklet.

This registration is for objective 1. Therefore, only details pertaining to that objective will be provided here.

ELIGIBILITY:
For physicians:

Inclusion criteria:

* age 18+
* working at an outpatient clinic in one of the participating hospitals.

Exclusion criteria:

* <18 years of age
* working at more than one of the participating hospitals

For patients:

Inclusion criteria:

* age 18+
* sought care at one of the outpatient clinics in the participating hospitals.

Exclusion criteria:

* <18 years of age
* one of the vulnerable populations (pregnant women, cognitively impaired adults)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2025-04-15 (Actual); Primary Completion 2025-11-28 (Actual); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Antibiotics prescription rate | 1-3 months before the intervention and 3-5 months after the intervention, depending on the timing of the intervention which varies by hospital.
  The number of patient visits in which antibiotics are prescribed by the total number of visits

SECONDARY OUTCOMES:
Differences in prescription rates by patient's gender | 1-3 months before the intervention and 3-5 months after the intervention, depending on the timing of the intervention which varies by hospital.
  The number of patient visits in which antibiotics are prescribed by the total number of visits, by male and female
Differences in prescription rates by patient's ethnicity (advantaged versus disadvantaged) | 1-3 months before the intervention and 3-5 months after the intervention, depending on the timing of the intervention which varies by hospital.
  The number of patient visits in which antibiotics are prescribed by the total number of visits, by advantaged and disadvantaged status

CONTACTS AND LOCATIONS:
Locations (2):
- Pennsylvania State University, University Park, Pennsylvania, United States
- Institute for Social and Environmental Research - Nepal, Bharatpur, Bagmati, Nepal

IPD SHARING:
Plan to Share IPD: No
There are potential risks about confidentiality, as the number of physicians is small.